CLINICAL TRIAL: NCT00904254
Title: The Use of Anti-CD4 mAb-Fragment for Imaging of Local Inflammation in Patients With Asymptomatic and Symptomatic Carotid Artery Stenosis - an Open Proof of Concept Study.
Brief Title: The Use of Anti-CD4 mAb-Fragment for Imaging of Local Inflammation in Patients With Carotid Artery Stenosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Technische Universität Dresden (Other)
Collaborators: Klinikum Chemnitz gGmbH (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TUD-Athero-040; 2008-008443-14 (EudraCT Number)
Record Dates: First submitted 2009-05-18; First posted 2009-05-19 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: Carotid Stenosis
Keywords: cerebrovascular disorders; symptomatic carotid artery stenosis; asymptomatic carotid artery stenosis; monoclonal antibody; diagnostics; molecular target; immunoglobulin Fab fragments; physiological effects of drugs; Tc99m-pertechnetate; Fab-fragment of Anti-human CD4; Antibodies, Monoclonal; Antibodies
MeSH Terms: conditions — Carotid Stenosis; Cerebrovascular Disorders | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1, diagnostic comparison (Experimental): EP 1645/Solution For Injection
  Interventions: Radiation: EP 1645/Solution For Injection, 99mTC

INTERVENTIONS:
Radiation: EP 1645/Solution For Injection, 99mTC — (Fab-fragment of Anti-human CD4,technetium-99m)
  Other Names: CD4 Antibody

SUMMARY:
The primary objective of this study is to proof the concept of EP 1645 as a diagnostic tool for carotid artery atherosclerosis and plaque instability and to assess the safety and tolerability of this diagnostic agent, a monoclonal antibody fragment (Fab') conjugated with the diagnostic radionuclide 99mTc. Safety and tolerability will be determined by adverse events (AEs) observed and reported upon administration of the product and the absorbed dose of radiation.

DETAILED DESCRIPTION:
For the evaluation of atherosclerosis in carotid arteries up to now sonographic measurements of plaque burden are used. This method has advantages for investigation of carotid arteries since this region is easy accessible for this investigation. However, it does not allow evaluation of the vessels which are remote from the body surface, as, for instance, coronary arteries. A method for non-invasive reliable evaluation of such arteries is needed. Also the distinction between vulnerable and stable plaque has a great clinical relevance. A quantifiable method for the determination of the effects of new therapeutic approaches would be highly appreciated.

It is expected, that the new antibody fragment with its radioactive linkage will allow displaying an image of the activity distribution of the disease. Due to the fact that only patients with atherosclerotic changes in carotid arteries allow comparing the activity and the clinical signs of disease, this proof of concept study (phase II study) will be performed in patients with asymptomatic and symptomatic carotid artery stenosis.

ELIGIBILITY:
Inclusion Criteria:

* male and female with either symptomatic (> 60%) or asymptomatic (> 80%) carotid artery stenosis between 50 and 80 years of age
* Symptomatic stenosis of the A. carotis interna is defined as occurence of focal ischemic symptoms in the area of the supplying vessel, occurence of a transischemic attack (TIA), occurence of focal neurologic dysfunction or unilateral blindness.
* informed consent in accordance with ICH GCP and § 40 AMG and StrahlSchV
* sonography status from the patient is present (printout is available)
* patients available for carotid surgery within 3 months after diagnosis of carotid artery stenosis
* In patients with bilateral disease, only the stenosis considered for surgery will be included in the endpoint evaluation.

Exclusion Criteria:

* patients > 80 years
* major disease of the cardiovascular system, respiratory system, hepatobiliary system or CNS, which prevents patients from the study participation as to the opinion of the investigator
* hepatic (transaminases > 3 x norm) or renal (serum creatinine increase > 2x norm) insufficiency
* regular drug intake of biologics. Intake of all other drugs must be judged by investigator and must be the strictly documented
* previous administration of xenogenous proteins
* history of anaphylactic reaction to any drug administered by a parenteral pathway
* previous participation in a radiopharmaceutical drug trial (unless the effective dose acquired by participation in the current trial will remain below 10 mSv)
* participation in any clinical drug trial within 3 months prior to enrolment
* women of child-bearing potential (child-bearing potential to be ruled out by one of the following: at least 2 years past menopause, hysterectomy, bilateral oophorectomy, bilateral tubal ligation)
* Patients presenting clinical signs of severe systemic infection (CRP > 50 mg/dl)
* Carotid Surgery (TEA) not possible within a time frame of 7 days after imaging
* Patients with bilateral carotid stenosis if clinically regarded as critical by the angiologists.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Scintigraphic confirmation of clinical disease | A total of 16 patients will be recruited for this study.
  8 patients with stable atherosclerosis will be assigned to study group 1 and 8 patients with instable atherosclerosis will be assigned to study group 2. It is expected that the study substance enriches only in carotid arteries of patients assigned to study group 2 and not in lesions of patients assigned to group 1. The study results of this proof-of-concept-study will be compared purely with descriptive methods in order to create a consistent set data which can be used for a valid case number estimation for a future phase II trial.

SECONDARY OUTCOMES:
Adverse events (signs and symptoms), laboratory tests. | during the entire study

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Schindler Schindler, MD, Principal Investigator — Institute of Clinical Pharmacology, Medical Faculty, Technical University Dresden